CLINICAL TRIAL: NCT03832504
Title: Identifying Optimal Cooling Strategies for Coronary Artery Disease Patients During Heatwaves
Brief Title: Identifying Strategies to Alleviate Cardiovascular Stress in Coronary Patients During Heatwaves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montreal Heart Institute (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Daniel Gagnon, Principal Investigator, Montreal Heart Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: ICM 2019-2425
Record Dates: First submitted 2019-01-21; First posted 2019-02-06 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — CCP110 protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 38°C and 60% RH + No intervention (Experimental): The participant will enter an environmental chamber maintained at 38°C and 60% relative humidity. The participant will remain within the environmental chamber and will rest in a seated position for 3 hours.
  Interventions: Other: No intervention
- 38°C and 60% RH + Fan (Experimental): The participant will enter an environmental chamber maintained at 38°C and 60% relative humidity. The participant will remain within the environmental chamber and will rest in a seated position for 3 hours.
  Interventions: Other: Fan
- 38°C and 60% RH + Skin wetting (Experimental): The participant will enter an environmental chamber maintained at 38°C and 60% relative humidity. The participant will remain within the environmental chamber and will rest in a seated position for 3 hours.
  Interventions: Other: Skin Wetting
- 38°C and 60% RH + Fan + Skin wetting (Experimental): Tthe participant will enter an environmental chamber maintained at 38°C and 60% relative humidity. The participant will remain within the environmental chamber and will rest in a seated position for 3 hours.
  Interventions: Other: Fan + Skin wetting
- 46°C and 10% RH + No intervention (Experimental): The participant will enter an environmental chamber maintained at 46°C and 10% relative humidity.
  Interventions: Other: No intervention
- 46°C and 10% RH + Skin wetting (Experimental): The participant will enter an environmental chamber maintained at 46°C and 10% relative humidity. The participant will remain within the environmental chamber and will rest in a seated position for 3 hours.
  Interventions: Other: Skin Wetting

INTERVENTIONS:
Other: No intervention — The participant will rest in a seated position.
  Arms: 38°C and 60% RH + No intervention; 46°C and 10% RH + No intervention
Other: Fan — A fan placed in front of the participant will provide an airflow of 4 m/s throughout the exposure.
  Arms: 38°C and 60% RH + Fan
Other: Skin Wetting — Tap water (~18°C) will be applied every 5 minutes to the face, neck, upper and lower arms and upper and lower legs using a spray bottle.
  Arms: 38°C and 60% RH + Skin wetting; 46°C and 10% RH + Skin wetting
Other: Fan + Skin wetting — A fan placed in front of the participant will provide an airflow of 4 m/s throughout the exposure. In addition, tap water (~18°C) will be applied every 5 minutes to the face, neck, upper and lower arms and upper and lower legs using a spray bottle.
  Arms: 38°C and 60% RH + Fan + Skin wetting

SUMMARY:
The purpose of this study is to determine the optimal cooling strategies to alleviate cardiovascular strain of coronary artery disease individuals during a simulated North American and Australian heatwave.

DETAILED DESCRIPTION:
Globally, heatwaves are occurring more frequently, are of greater intensity and longer in duration. The devastating health impacts of extreme heat are increasingly recognized, particularly in vulnerable populations, such as adults with coronary artery disease (CAD). While the most effective cooling strategy during a heatwave is the use of air conditioning (AC), economical concerns can limit AC use among vulnerable populations. In addition, widespread AC use places a significant burden on the electrical grid, causing brown-outs and black-outs during periods of extreme heat.

Electric fans offer a cooling strategy with a 50-fold lower power requirement and cost compared to AC. However, the efficacy of fan use during heat waves remains contentious. The primary objective of this study is to identify the optimal cooling strategy to alleviate cardiovascular strain of CAD patients exposed to typical North American heatwave conditions (38°C with 60% relative humidity). The secondary objective is to identify the optimal cooling strategy to alleviate cardiovascular strain of CAD patients exposed to typical Australian heatwave conditions (46°C with 10% relative humidity).

ELIGIBILITY:
Inclusion Criteria:

* History of angiographic coronary disease (≥70% arterial diameter narrowing of at least one major epicardial coronary artery) and/or prior coronary revascularization and/or documented prior acute coronary syndrome and/or stable angina and/or perfusion defect during exercise testing.
* No CAD-related hospitalisations or changes in cardiac medications or change in pattern of angina for at least 3 months prior to enrolment

Exclusion Criteria:

* Body mass index ≥35 kg/m2.
* Currently undertaking estrogen therapy.
* Evidence of current fluid and electrolyte disorders, anemia, abnormal thyroid function, arrhythmias, diabetes, renal disease, liver disease, cerebrovascular disease, significant pulmonary disease, endocrine abnormalities, significant cognitive impairment, psychiatric disorder, substance abuse, degenerative neurological condition or any other medical condition deemed to pose risk during the proposed experiments.
* Uncontrolled hypertension (>180/110 mmHg).
* Recent (<3 months) coronary bypass surgery.
* Ejection fraction <40% and/or clinical evidence/history of heart failure.
* Significant valvular heart disease
* Resting ECG abnormalities interfering with observation of ST segment changes during testing.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Rate pressure product | Change from baseline to the end of the 3 hour exposure
  Rate pressure product, in beats per minute per mmHg

SECONDARY OUTCOMES:
Body core temperature | Change from baseline to the end of the 3 hour exposure
  In degrees Celcius

OTHER OUTCOMES:
Skin temperature | Change from baseline to the end of the 3 hour exposure
  In degrees Celcius
Sweat loss | Change from baseline to the end of the 3 hour exposure
  In kilograms
Local sweat rate | Measured continously during the 3 hour exposure
  In mg per minute per cm2
Skin blood flow | Measured continously during the 3 hour exposure.
  In arbitrary perfusion units

CONTACTS AND LOCATIONS:
Locations (1):
- cardiovascular Prevention and rehabilitation Centre of the Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
All individual data will be de-identified and available to the public through publications, media articles and conference presentations